CLINICAL TRIAL: NCT04911647
Title: A Prospective Randomized Multi-center Study for Efficacy of Metallic Biliary Stent Compared to Plastic Stent in Patients Receiving Neoadjuvant Chemotherapy for Resectable Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0115
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Resectable Pancreatic Cancer With Biliary Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Plastic stent (Active Comparator): Patient group with plastic stent inserted in biliary obstruction through endoscope
  Interventions: Device: ERCP using plastic stent
- The metal stent (Experimental): Patient group with metal stent inserted in biliary obstruction through endoscope
  Interventions: Device: ERCP using metal stent

INTERVENTIONS:
Device: ERCP using plastic stent — Insertion of plastic stent (plastic stent with inner diameter 1.8mm or more) in the biliary obstruction will be performed using ERCP in the patients with the pancreatic cancer undergoing neoadjuvant therapy.
  Arms: The Plastic stent
Device: ERCP using metal stent — Insertion of metal stent (full covered self-expandable metal stent) in the biliary obstruction will be performed using ERCP in the patients with the pancreatic cancer undergoing neoadjuvant therapy.
  Arms: The metal stent

SUMMARY:
Pancreatic cancer is the eighth most common occurrence in Korea. In the United States, pancreatic cancer is expected to be the number two cause of death from cancer in 2030. The prevalence of pancreatic cancer is also on the rise in Korea. The 5-year survival rate of pancreatic cancer in Korea is 10.8%. According to the 2017 cause of death statistics, pancreatic cancer mortality is ranked fifth. It is known to have the worst prognosis of cancer in the body. The median survival period of unresectable pancreatic cancer is only six months, and resection is the only treatment that can be expected to be completely cured, but only about 10% of cases are possible to be operable at the time of diagnosis.

In the 2000s, the studies began to emerge on diagnosis and treatment of pancreatic cancer with intermediate anatomical and imaging characteristics of resectable and locally advanced pancreatic cancer. Margin negative resection plays an important role in the long-term survival rate in surgical treatment of pancreatic cancer. Prior to 2001, pancreatic cancer with invasion of vein was considered impossible to perform radical resection. However, the studies have been published that a satisfactory long-term survival rate and margin negative resection could be obtained when venous resection was performed along with radical resection. Since the 2006, the National Comprehensive Cancer Network (NCCN) guideline, after performing radical resection among locally advanced pancreatic cancers without remote metastasis, pancreatic cancers with high risk of margin positive resection and treatment failure were classified as "borderline resectable". In the borderline resectable pancreatic cancer, neoadjuvant therapy was recommended before surgery. In recent years, the neoadjuvant therapy has been reported to raise the survival rate in resectable pancreatic cancer. Furthermore, a prospective study is in progress to demonstrate the effectiveness of neoadjuvant therapy with FOLFIRINOX in resectable pancreatic cancer. If pancreatic cancer is located in the head of pancreas, jaundice can be occurred often. In the case of preoperative jaundice, the possibility of postoperative complications increases. So biliary drainage is performed before surgery. In biliary drainage, usually the plastic stent was inserted through the endoscope. If the metal stent is inserted in the biliary obstruction, it can cause severe inflammation around the bile duct due to the radial force, and it is difficult to remove in the surgery. However, the meta-analysis comparing the groups of metal and plastic stents in the recent preoperative biliary drainage showed no difference of postoperative complication, and postoperative pancreatic fistula was lower in the group of metal stents (5.1% vs. 11.8% p=0.04). In addition, fewer re-intervention cases before surgery were found in the group of metal stents (3.4% vs.14.8% p < 0.0001).

Not only in the borderline resectable, but also in the resectable pancreatic cancer, neoadjuvant therapy has recently been actively performed in the cases of large tumor size, high CA 19-9, large lymph nodes, severe weight loss, and severe pain. The comparison study of the efficacy between plastic and metal stents in preoperative bile drainage in pancreatic cancer with neoadjuvant therapy has not yet been prospectively performed. However, retrospective studies have shown that metal stents have a lower re-treatment rate than plastic stent (0.24 vs 0.54), and that there is no difference in post-operative complications. Therefore, we planned the study to compare the efficacy and safety between metal and plastic stent in biliary drainage performed in patients undergoing neoadjuvant therapy with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 years or older who have confirmed histologically or radiologically resectable pancreatic cancer
2. Patients with clinical obstruction symptoms and radiographically confirmed biliary obstruction related to malignant tumors
3. Patients receiving neoadjuvant chemotherapy before surgery

Exclusion Criteria:

1. Patients diagnosed as unresectable pancreatic cancer
2. Patients with biliary obstruction due to biliary cancer, not pancreatic cancer
3. Patients with duodenal obstruction
4. Patients with pancreatic cance and other cancers
5. Patients with severe uncontrolled infection
6. Patients with 3 or higher of performance score as the Eastern Cooperative Oncology Group
7. Patients who have not agreed with the informed consent
8. Patients who are technically unable to be undergone endoscopic procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Re-intervention rate | 6 months
  Re-intervention because of obstructive jaundice, cholangitis, stent malfunction, complication of procedure of ERCP

SECONDARY OUTCOMES:
Procedure related complication, Postoperative complication | 6 months
  1. Complication because of procedure (ERCP)
  2. Complication because of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Seung Min Bang, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No